CLINICAL TRIAL: NCT07209878
Title: 68Ga-PSMA-11 PET Imaging in the Diagnostic Study of Newly Diagnosed, Untreated Prostate Cancer, With a Head-to-head Comparison to mpMRI
Brief Title: 68Ga-PSMA-11 PET Imaging for Diagnosing Prostate Cancer, a Head-to-head Comparison With mpMRI
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-68Ga-PSMA-11
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: PSMA; Prostate cancer; PET imaging; mpMRI
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA-11 PET/CT (Experimental): Intravenous injection of 68Ga-PSMA-11 with a dosage of 111-148 MBq (3-4 mCi), followed by PET/CT or PET/MRI acquisition according to standard methods
  Interventions: Drug: 68Ga-PSMA-11

INTERVENTIONS:
Drug: 68Ga-PSMA-11 — Intravenous injection of 68Ga-PSMA-11 with a dosage of 111-148 MBq (3-4 mCi), followed by PET/CT or PET/MRI acquisition according to standard methods.

SUMMARY:
68Ga-PSMA-11 is a widely used radiotracer targeting PSMA. In this study, we investigated the diagnostic efficacy of 68Ga-PSMA-11 PET imaging (PET/CT or PET/MRI) in patients with newly diagnosed, treatment-naive prostate cancer, and performed a head-to-head comparison with multi-parameter magnetic resonance imaging (mpMRI).

DETAILED DESCRIPTION:
68Ga-PSMA-11 is a radiotracer targeting PSMA. Previously, multiple clinical trials have validated the clinical applications of 68Ga-PSMA-11 PET. Meanwhile, multi-parametric magnetic resonance imaging (mpMRI) still holds a dominant position in the imaging diagnosis of prostate cancer. In this study, we will further evaluate the diagnostic performance of 68Ga-PSMA-11 positron emission tomography (PET/CT or PET/MRI) in newly diagnosed and untreated prostate cancer patients, with a head-to-head comparison to mpMRI.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed adenocarcinoma of the prostate.
* No anti-tumor treatment received prior to the PET imaging.
* Subjects provide signed informed consent and confirm that they are able and willing to comply with all protocol requirements.
* Radical prostatectomy scheduled within 28 days after PET imaging

Exclusion Criteria:

* Patients with other malignant tumors
* Subjects with any medical condition or other circumstance that, in the opinion of the investigator, compromise obtaining reliable data, achieving study objectives, or completion.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of 68Ga-PSMA-11 Imaging to Detect Intraprostatic Tumors Relative to Histopathology in newly diagnosed, treatment-naive Prostate Cacner Participants | Within 28 days of imaging, radical prostatectomy will occur.
  Using histopathology from radical prostatectomy as the reference standard, validate the true positive detection rate of PET for prostate lesions. Two experienced nuclear medicine physicians, blinded to all other imaging and clinical history of the patients, independently assessed the PET images. Any disagreements were resolved by consensus.
Specificity of 68Ga-PSMA-11 PET Imaging to Detect Intraprostatic Tumors Relative to Histopathology in newly diagnosed, treatment-naive Prostate Cacner Participants | Within 28 days of imaging, radical prostatectomy will occur.
  Using histopathology from radical prostatectomy as the reference standard, validate the true negative detection rate of PET for prostate lesions. Two experienced nuclear medicine physicians, blinded to all other imaging and clinical history of the patients, independently assessed the PET images. Any disagreements were resolved by consensus.

SECONDARY OUTCOMES:
Comparison of Detection Rates for Intraprostatic Tumors Between 68Ga-PSMA-11 PET Imaging and mpMRI | Within 1-2 hours of 68Ga-PSMA-11 dosing, a whole body PET scan will be taken
  The number of intraprostatic lesions detected on imaging will be determined by each of independent readers. The sum of lesions per participant per tissue type and overall will be computed for each participant based on each reader's lesion count. This will be calculated from the 68Ga-PSMA-11 PET scan results as well as the mpMRI results.

CONTACTS AND LOCATIONS:
Overall Officials: Weibign Miao, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China